CLINICAL TRIAL: NCT06641661
Title: The Association Between NPC1L1 Gene Polymorphism and the Efficacy and Safety of Hybutimibe in High/very High Risk ASCVD Patients
Brief Title: NPC1L1 Gene Polymorphism and the Efficacy and Safety of Hybutimibe
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Beijing Micro Love Public Welfare Foundation (Unknown)
Responsible Party: Principal Investigator, Mei Gao, Clinical Professor, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2024（067)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Gene Polymorphism; ASCVD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental group: Hybutimibe 10mg QD was added to the conventional treatment
  Interventions: Drug: Hybutimibe 10mg QD

INTERVENTIONS:
Drug: Hybutimibe 10mg QD — Hybutimibe was added to the conventional treatment

SUMMARY:
Significant individual differences may lead to differences in patients' responses to drug therapy and lead to an increased incidence of adverse reactions. However, there are currently very limited data on the genetic variation of the NPC1L1 gene in the Chinese population. In view of the important role of NPC1L1 gene polymorphism in cholesterol absorption, lipid profile, coronary heart disease prevalence and ezetimibe response, it is necessary to focus on the allele frequency analysis of NPC1L1 gene polymorphism in the Chinese population, and to further explore the therapeutic response of NPC1L1 gene polymorphism and Hybutimibe.

With reference to previous domestic and foreign literature reports and HapMap project (http://hapmap.ncbi.nlm. nih.gov/)SNP) distribution, this study selected NPC1L1 gene loci with relatively in-depth clinical research. rs2072183, rs4720470, rs2073547 were analyzed. The minimum allele frequency (MAF) of the above loci were all greater than 10%, and it has been confirmed that genetic variation exists between different diseases and different races, which may affect the lipid profile , the risk of coronary heart disease and the response to hybomaib treatment. However, the variability of rs2072183 in response to Hybutimibe needs to be further verified, and the effects of rs4720470 and rs2073547 gene polymorphisms on drug response also need to be targeted. In order to further determine the correlation between the distribution of NPC1L1 polymorphism and the efficacy and safety of Hybutimibe, we conducted this study to observe the distribution frequency of NPC1L1 gene polymorphisms at rs2072183, rs4720470 and rs2073547 in high-risk/extremely high-risk ASCVD patients. To explore the correlation between NPC1L1 gene polymorphisms and the efficacy and safety of Hybutimibe combined with moderate-intensity statins in the treatment of high-risk/very high-risk ASCVD patients. This is the first time to explore the distribution of NPC1L1 polymorphism in high/very high risk ASCVD population in China, which will provide genetic evidence for the correct use of Hybutimibe and moderate intensity statin therapy, and provide further evidence-based medical evidence for the distribution of NPC1L1 polymorphism and the efficacy and safety of Hybutimibe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high/very high risk of ASCVD were only treated with moderate intensity statins (including atorvastatin 10-20mg, rosuvastatin 5-10mg, fluvastatin 80mg, lovastatin 40mg, pivastatin 1-4mg, pravastatin 40mg, simvastatin 20-40mg, etc.) for at least 8 weeks before enlistment.
2. The LDL-C level did not meet the lipid reduction target corresponding to the risk stratification level of ASCVD recommended by the Chinese Lipid Management Guidelines (2023), or the level of LDL-C was still not up to the standard as clinicians expected that patients should continue to use medium-dose statins for lipid-lowering treatment alone, and the cholesterol absorption inhibitor Hybomab should be combined;
3. Age 18-75 years old;
4. BMI range 22-45 kg/m2;
5. Can understand and voluntarily sign informed consent.

Exclusion Criteria:

1. Allergic history of cholesterol absorption inhibitors and statins;
2. other types of cholesterol absorption inhibitors have been used;
3. Homozygous familial hypercholesterolemia;
4. any clinically serious endocrine disease affecting blood lipids or lipid proteins;
5. Abnormal liver function with AST or ALT greater than three times the upper limit of normal, or bilirubin >34uM, creatine muscle enzyme greater than five times the upper limit of normal, or evidence of serologically infectious liver disease;
6. Thyroid dysfunction;
7. History of malignant tumor;
8. Patients with coagulation dysfunction;
9. Women who are pregnant or planning to become pregnant;
10. Taking fenofibrate, gefilozil, probucol, warfarin, glucocorticoids, cyclosporine or another immunosuppressant within 30 days prior to the trial;
11. can not adhere to medication or regular follow-up;
12. Communication disorders, people with severe aphasia, audio-visual impairment, serious mental illness, and difficulty cooperating with investigators;
13. There are other circumstances that the researcher considers inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high/very high risk of ASCVD who were treated with only moderate-intensity statins for at least 8 weeks before enlistment and whose LDL-C levels did not meet the lipid reduction target corresponding to the risk stratification level of ASCVD recommended by the Chinese Lipid Management Guidelines (2023) and who needed to be combined with Hybutimibe.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of LDL-C change from baseline at week 12 of treatment | at week 12 of treatment
  Rate of LDL-C change from baseline in high-risk/very high-risk ASCVD patients at week 12 of treatment

SECONDARY OUTCOMES:
At the 4th week of treatment, LDL-C change rate from baseline in high-risk/very high-risk ASCVD patients | At the 4th week of treatment
  At the 4th week of treatment, LDL-C change rate from baseline in high-risk/very high-risk ASCVD patients
Changes in HDL-C, TC and TG levels at the 4th and 12th week of treatment. | at the 4th and 12th week of treatment
  Changes in HDL-C, TC and TG levels at the 4th and 12th week of treatment.
Changes in levels of alanine aminotransferase, aspartate aminotransferase and creatine kinase at the 4th and 12th week of treatment. | at the 4th and 12th week of treatment
  Changes in levels of alanine aminotransferase, aspartate aminotransferase and creatine kinase at the 4th and 12th week of treatment.
Polymorphism and distribution frequency of NPC1L1 gene rs2072183, rs4720470 and rs2073547 in high-risk/extremely high-risk ASCVD patients. | at enrollment
  Polymorphism and distribution frequency of NPC1L1 gene rs2072183, rs4720470 and rs2073547 in high-risk/extremely high-risk ASCVD patients.

CONTACTS AND LOCATIONS:
Overall Officials: mei Gao, Doctor, Study Chair — Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No